CLINICAL TRIAL: NCT03408912
Title: CMR or Angiography for FFR-guided Revascularisation in ST-elevation Myocardial Infarction
Brief Title: CMR or Angiography for FFR-guided Revascularisation
Acronym: CRAFT-MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Martin Ugander, MD, PhD, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/1821-31
Record Dates: First submitted 2017-12-19; First posted 2018-01-24 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMR and angiography FFR (Other): Patients will undergo both CMR and angiography to acquired FFR.
  Interventions: Diagnostic Test: FFR

INTERVENTIONS:
Diagnostic Test: FFR — FFR from CMR compared to invasive FFR

SUMMARY:
Around 50% of patients that present with ST Elevation Myocardial Infarction (STEMI) have residual disease in the non-culprit lesions. If the residual disease should be treated, what should guide intervention? Fractional Flow Reserve (FFR) has been proposed as a guide for intervention, however new developments in cardiovascular magnetic resonance (CMR) allows for non-invasive FFR measurements.

If FFR from CMR can predict physiological significant stenosis as good as FFR from invasive angiography, unnecessary invasive producers can be avoided in patients with STEMI.

DETAILED DESCRIPTION:
Early reperfusion of epicardial coronaries is essential for salvage of ischemic myocardium, reducing both morbidity and mortality in patients with ST elevation myocardial infarction (STEMI). Current European Society of Cardiology guidelines recommend percutaneous coronary intervention (PCI) of the infarct related artery (IRA) for patients presenting with STEMI, with residual disease initially being treated conservatively. Large meta-analyses of observational studies have shown that PCI of the IRA only results in a reduced mortality compared to full revascularization in patients with STEMI and simultaneous multivessel disease. However, recent small randomized controlled trials indicate that full revascularization reduces morbidity, but have been underpowered to show any reduction in mortality. Furthermore, physiological guidance of coronary intervention by fractional flow reserve (FFR) reduces mortality compared to angiography guided PCI in both stable angina and non-STEMI (NSTEMI). However, if performing full revascularization guided by FFR in patients with STEMI improves clinical outcome, compared to initial conservative approach is not known.

Assessment of myocardial perfusion in rest and during pharmacological stress is widely used for non-invasive diagnosis of myocardial ischemia, where cardiovascular magnetic resonance (CMR) has a high diagnostic accuracy. Newly developed first pass perfusion imaging with cardiovascular magnetic resonance (CMR) allows for quantification of myocardial perfusion, and CMR derived FFR. However, it is currently not known if FFR from CMR and invasive angiography correlate with each other. If FFR from CMR can predict physiological significant stenosis as good as FFR from invasive angiography, unnecessary invasive producers can be avoided in patients with STEMI.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the active arm of FULL REVASC, that has not undergone invasive FFR, and give written informed consent.

Exclusion Criteria:

* Asthma/Chronic Obstructive Pulmonary Disease, systolic blood pressure under 90 mmHg, bradycardia (less than 45 beats/min), persistent second or third AtrioVentricular-block, Sick Sinus Syndrome, Long QT Syndrome, atrial fibrillation, severe aortic stenosis, severe heart failure (NHYA class III-IV), metallic implants, kidney failure (less than 30 ml/min/1.73 square meters body surface area), current treatment with the drugs Persantin, theophyllamin or Fevarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The agreement between CMR-derived FFR and FFR from angiography | Measurements will be collected within 1-2 days of each other.
  FFR will be measured with CMR on day one. FFR will be measured with invasive angiography on the following day. The FFR acquired with both methods will be compared with Pearson's correlation coefficient and Bland-Altman analysis. The aim of the study is to validate the agreement between CMR-derived FFR with FFR from angiography as the independent reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ugander, MD, PhD, Principal Investigator — Karolinska Institutet; Felix Böhm, MD, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No